CLINICAL TRIAL: NCT00689663
Title: Randomized Multicentre Trial: Comparison of Harmonic Ace and Eletrocautery; Comparison of Fundus First and Conventional Dissection
Brief Title: Laparoscopic Cholecystectomy - Fundus First and Harmonic Ace Compared With Conventional Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sundsvall Hospital (Other)
Responsible Party: Divisionschef Margaretha Röden, Landstinget Västernorrland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YC11
Record Dates: First submitted 2008-05-26; First posted 2008-06-03 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2008-05

CONDITIONS: Cholecystectomy
Keywords: cholecystectomy
MeSH Terms: interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Dissection staring at the triangle of calots. Dissection with electrocautery.
  Interventions: Procedure: Laparoscopic cholecystectomy
- 2 (Active Comparator): Dissection as fundus first with electrocautery.
  Interventions: Procedure: Laparoscopic cholecystectomy
- 3 (Active Comparator): Dissection as fundus first with ultrasonic dissection.
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Randomized to three arm.
  Other Names: Randomised study.

SUMMARY:
Laparoscopic cholecytectomy can be by starting the dissection at the triangle of calots or as a fundus first dissection.

Dissection can be with electrocutery or ultrasonic. The optimal technique or the optimal way of dissection has to be established. Patients are at 4 hospitals randomised to the different techniques and the different methods of dissection.

DETAILED DESCRIPTION:
Patients at the participating hospitals are randomized to:

1. dissection starting at the triangle of Calots with electrocautery.
2. dissection by fundus first technique with electrocautery.
3. dissection by fundus first technique with ultrasonic dissection.

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic cholecystectomy

Exclusion Criteria:

* age >Z65
* ASA >3
* obesity
* previous extensive gastrointestinal surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2006-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Operation time, bleeding, pain, nausea, quality of life, analgetics, sick leave, surgical complications, conversion rate | 30 days

SECONDARY OUTCOMES:
surgical complications | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Leif A Israelsson, MD,PhD, Study Chair — Umea University
Locations (1):
- Sundsvall Hospital, Sundsvall, Sundsvall, Sweden

REFERENCES:
- [Background] Cengiz Y, Janes A, Grehn A, Israelsson LA. Randomized trial of traditional dissection with electrocautery versus ultrasonic fundus-first dissection in patients undergoing laparoscopic cholecystectomy. Br J Surg. 2005 Jul;92(7):810-3. doi: 10.1002/bjs.4982. PMID 15880649